CLINICAL TRIAL: NCT05901974
Title: A Multicenter Prospective Clinical Study of Venetoclax Combined With Azactidine in the Treatment of Acute Leukaemias of Ambiguous Lineage
Brief Title: Venetoclax Combined With Azactidine in the Treatment of ALAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheng-Li Xue, MD (Other)
Collaborators: Jining Medical University (Other); The Second People's Hospital of Huai'an (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Affiliated Hospital of Nantong University (Other); Suzhou Hospital of Traditional Chinese Medicine (Other); Northern Jiangsu People's Hospital (Other); Pingdingshan first people's Hospital (Unknown); The Second Affiliated Hospital of Wannan Medical College (Unknown); Canglang Hospital of Suzhou (Unknown)
Responsible Party: Sponsor-Investigator, Sheng-Li Xue, MD, Professor, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZALAL01
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Leukemia of Ambiguous Lineage
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax Combined With azactidine in the Treatment of Acute Leukaemias of Ambiguous Lineage (Experimental): Venetoclax combined with azacitidine regimen. Venetoclax orally once daily (100 mg d1, 200 mg d2, 400 mg d3-28); azacitidine 75 mg/m2 subcutaneously once daily on days 1-7 .
  Interventions: Drug: Venetoclax; Drug: azactidine

INTERVENTIONS:
Drug: Venetoclax — Venetoclax orally once daily (100 mg d1, 200 mg d2, 400 mg d3-28);
Drug: azactidine — azacitidine 75 mg/m2 subcutaneously once daily on days 1-7

SUMMARY:
The prognosis of acute leukaemias of ambiguous lineage is poor. The effect of chemotherapy regimen and hematopoietic stem cell transplantation are still unclear. Therefore, we will explore new therapy to improve the remission rate of acute leukaemias of ambiguous lineage. Venetoclax can significantly improve the remission rate and prolong PFS and OS. At present, venetoclax combined with azacitidine or decitabine has become the preferred treatment regimen for elderly AML patients. It also shows a high response rate in relapsed/refractory AML or MDS patients. There are few clinical studies on the treatment of ALAL. The purpose of this study is to explore the efficacy and safety of venetoclax combined with azacitidine in the treatment of newly diagnosed ALAL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 15 years.
2. Patients diagnosed with ALAL according to 5th edition of WHO Acute Leukaemias of Ambiguous Lineage diagnosis standard.
3. New diagnosed patients.
4. ECOG performance status score less than 3.
5. Expected survival time ≥3 months.
6. Patients without serious heart, lung, liver, or kidney disease.
7. Ability to understand and voluntarily provide informed consent.

Exclusion Criteria:

1. Patients who are allergic to the study drug or drugs with similar chemical structures.
2. Pregnant or lactating women, and women of childbearing age who do not want to practice effective methods of contraception.
3. Active infection.
4. Active bleeding.
5. Patients with new thrombosis, embolism, cerebral hemorrhage, or other diseases or a medical history within one year before enrollment.
6. Patients with mental disorders or other conditions whereby informed consent cannot be obtained and where the requirements of the study treatment and procedures cannot be met.
7. Liver function abnormalities (total bilirubin > 1.5 times the upper limit of the normal range, ALT/AST > 2.5 times the upper limit of the normal range or patients with liver involvement whose ALT/AST > 1.5 times the upper limit of the normal range), or renal anomalies (serum creatinine > 1.5 times the upper limit of the normal value).
8. Patients with a history of clinically significant QTc interval prolongation (male > 450 ms; female > 470 ms), ventricular heart tachycardia and atrial fibrillation, II-degree heart block, myocardial infarction attack within one year before enrollment, and congestive heart failure, and patients with coronary heart disease who have clinical symptoms and requiring drug treatment.
9. Surgery on the main organs within the past six weeks.
10. Drug abuse or long-term alcohol abuse that would affect the evaluation results.
11. Patients who have received organ transplants (excepting bone marrow transplantation).
12. Patients not suitable for the study according to the investigator's assessment.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | At the end of Cycle 1 (each cycle is 28 days)
  The overall response (complete remission, complete remission with incomplete blood count recovery) rate achieved after one or two courses (28 days) induction therapy by venetoclax combined azacitidine regimen.
Complete Remission Rate (CRR) | At the end of Cycle 1 (each cycle is 28 days)
  The complete remission rate achieved after one or two courses (28 days) induction therapy by venetoclax combined azacitidine regimen.

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year
  It is measured from the date of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Progression-Free Survival (PFS) | 1 year
  It is measured from the date of entry into this trial to the date of progression or death.
Adverse events in hematological system | 1 year
  Record of adverse events in hematological system during and after designed venetoclax combined azacitidine regimen induction.
Adverse events in other organs or systems | 1 year
  Record of adverse events in other organs or systems during and after designed venetoclax combined azacitidine regimen induction.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No